CLINICAL TRIAL: NCT01711177
Title: Effect of Travoprost 0.004% on Retinal Oximetry in Primary Open Angle Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Pierre Forcier, Associate professor, Université de Montréal
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPM3117-Dubois/Pham
Record Dates: First submitted 2012-10-03; First posted 2012-10-22 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-06

CONDITIONS: Primary Open Angle Glaucoma
Keywords: primary open angle glaucoma; retinal oximetry
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Travoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Normal control (Sham Comparator): Normal patient placebo
  Interventions: Drug: placebo
- Glaucoma suspect (Sham Comparator): Patients with elevated Intraocular pressure higher than 18 mmHg (placebo)
  Interventions: Drug: placebo
- Newly diagnosed glaucoma (Experimental): Treated with Travoprost (0.04%)
  Interventions: Drug: travoprost

INTERVENTIONS:
Drug: placebo — Placebo
  Arms: Glaucoma suspect; Normal control
Drug: travoprost — Travatan Z is administered to newly diagnosed glaucoma patient
  Other Names: travatan
  Arms: Newly diagnosed glaucoma

SUMMARY:
Glaucoma is the second leading cause of blindness among seniors in Canada. It is often associated with an elevated intraocular pressure (IOP), but its exact mechanism is still largely unknown. Some studies have shown a link between glaucoma and changes in the amount of oxygen in the veins of the eye. The study aims to compare the amount of oxygen in ocular veins among three different groups using a spectrophotometer. This instrument is linked to a camera and can measure the quantity of oxygen in the veins using different characteristics of the blood inside.

The groups of the study are: patients without glaucoma, patients suspected of glaucoma and patients newly diagnosed with glaucoma. The drug the investigators are using, Travoprost 0.004%, will only be administered to the groups suspected or diagnosed with glaucoma. Travoprost 0.004% is already approved for use in Quebec and is part of standard care. Ten patients will be recruited into each group for a total of 30 patients in this study. All patients for the suspected or diagnosed groups will be recruited from the Jewish General Hospital. Subsequently all testing will be done at the École d'optométrie, Université de Montréal

ELIGIBILITY:
Inclusion Criteria:

* good systemic health
* irido-corneal angle open
* intraocular pressure more than 18 mmHg

Exclusion Criteria:

* having cardiovascular problem
* Hypertension or diabetes
* under systemic medication for high blood pressure
* had an ocular surgery in the past

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Montreal, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Normal Control | Glaucoma Suspect | Newly Diagnosed Glaucoma
Started | 10 | 3 | 3
Completed | 10 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Control | Glaucoma Suspect | Newly Diagnosed Glaucoma | Total
Number analyzed (Participants) | 10 | 3 | 3 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 3 | 2 | 15
  >=65 years | 0 | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (5) | 53 (8) | 60 (9) | 55 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 9
  Male | 5 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Blood Oxygenation
Description: For each subject, all the measurements will be done during an 1 hour appointment.
Time Frame: 1 hour
Measure: Mean (95% Confidence Interval); unit: percentage of oxygenation
Arm/Group | Normal Control | Glaucoma Suspect | Newly Diagnosed Glaucoma
Number analyzed (Participants) | 10 | 3 | 3
percentage of oxygenation | 60 [55 to 63] | 60 [55 to 63] | 60 [55 to 63]

ADVERSE EVENTS:
Time Frame: 6 month
Arm/Group | Normal Control | Glaucoma Suspect | Newly Diagnosed Glaucoma
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/10 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes